CLINICAL TRIAL: NCT06197893
Title: Comparison of Conventional and Modified Sling Suture Techniques In Free Gingival Graft Operations With CAIRO Type 2 and Type 3 Localized Gingival Recessions
Brief Title: Modified Sling and Conventional Suture Techniques in Free Gingival Graft Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Sanubar Shakiliyeva, Periodontology specialist, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSHAKILIYEVA
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Gingival Recession, Localized
Keywords: Gingival unit graft; Sling suture; Shrinkage
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. GUG+MSS (Experimental): The GUG was obtained from the maxillary premolar area. The dissected graft was fixed to the recipient site using a modified sling suture technique.
  Interventions: Procedure: gingival unit graft+modified sling suture technique
- 2. GUG+CS (Experimental): The GUG was obtained from the maxillary premolar area, as detailed experimental GUG+MSS group. The dissected graft was fixed to the recipient site using conventional suture technique.
  Interventions: Procedure: Gingival unit graft and conventional suture technique
- 3. CG+MSS (Experimental): Conventional graft dimensions were determined with aluminum foil and the foil was placed in the palatial region at the level of the maxillary premolars, at least 2 mm away from the free gingival margin of the adjacent teeth. The dissected graft was fixed to the recipient site with 5/0 polypropylene suture using a modified sling suture technique, as detailed experimental GUG+MSS group.
  Interventions: Procedure: Conventional graft and modified sling suture technique
- 4. CG+CS (Experimental): The dissected conventional graft, as detailed experimental CS+MSS group, fixed recipient bed with conventional suture technique, as detailed experimental GUG+CS group.
  Interventions: Procedure: Conventional graft and conventional suture technique

INTERVENTIONS:
Procedure: gingival unit graft+modified sling suture technique — The GUG was obtained from the maxillary premolar area. A sulcular incision including the marginal gingival tissue, and two vertical incisions, including the distal and mesial papillae, was made in the palatial parts of the premolars. Then, the incision lines were combined and a 1-1.5 mm thick graft of the desired dimensions was dissected. The dissected graft was fixed to the recipient site with 5/0 polypropylene suture using a modified sling suture technique. First, the needle was passed through the graft slightly apical to the mesial papilla on the buccal side and removed from the lingual aspect including lingual papilla. Subsequently, on the distal side, the needle was passed from the lingual side to the buccal side, and it was passed through the graft slightly apical to the distal papilla and removed from the lingual gingiva again. Then it was knotted on the buccal graft by returning to the buccal starting point on the mesial side.
  Arms: 1. GUG+MSS
Procedure: Gingival unit graft and conventional suture technique — The GUG was obtained from the maxillary premolar area. The dissected graft was fixed to the recipient site with 5/0 polypropylene suture using conventional suture technique. Conventional suture technique includes a horizontal matrix suture and 2 simple sutures. First the coronal part of the dissected graft was fixed to the recipient bed with a horizontal matrix suture, then with 2 simple sutures along the vertical incision line from mesial and distal sides with 5/0 polypropylene suture.
  Arms: 2. GUG+CS
Procedure: Conventional graft and modified sling suture technique — Conventional graft dimensions were determined with aluminum foil and the foil was placed in the palatinal region at the level of the maxillary premolars, at least 2 mm away from the free gingival margin of the adjacent teeth. The exterier edges of the foil were drawn with a scalpel and the 1-1.5 mm thick graft was dissected from the donor site. The dissected graft was fixed to the recipient site with 5/0 polypropylene suture using a modified sling suture technique.
  Arms: 3. CG+MSS
Procedure: Conventional graft and conventional suture technique — Conventional graft obtained from the palatinal region at the level of the maxillary premolars, at least 2 mm away from the free gingival margin of the adjacent teeth. The dissected graft was fixed to the recipient site with 5/0 polypropylene suture using conventional suture technique.
  Arms: 4. CG+CS

SUMMARY:
The aim of this study is to investigate the effects of conventional suture (CS) and modified sling suture (MSS) techniques, applied in free gingival graft (FGG) surgery using gingival unit graft (GUG) and conventional graft (CG) techniques, on clinical parameters and graft dimensions.

DETAILED DESCRIPTION:
Background: The aim of this study is to investigate the effects of conventional suture (CS) and modified sling suture (MSS) techniques, applied in free gingival graft (FGG) surgery using gingival unit graft (GUG) and conventional graft (CG) techniques, on clinical parameters and graft dimensions.

METHODS: 52 individuals having Cairo Type 2 (RT2) and Type 3 (RT3) gingival recessions in mandibular anterior region were divided into four groups as a) GUG+MSS (n=13), b) GUG+CS (n=13), c) CG+MSS (n=13) and d) CG+CS (n=13). Keratinized gingival width (KGW), keratinized tissue thickness (KGT), relative gingival recession height (rGRH), and relative vestibule depth (rVD) measurements were recorded using a digital caliper and periodontal probe UNC 15. Dimensional changes (Δ) of the graft surface area (GSA) was determined by ImageJ software. All measurements were done at baseline and repeated 1st and 3rd months.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals
* <1 mm of attached gingiva on mandibular incisors
* PI and GI scores <1
* Patients who had not previously undergone soft tissue surgery in the relevant area

Exclusion Criteria:

* Pregnant or lactating women
* Patients younger than 18 years old
* Mandibular incisors with having restoration, probing depth ≥ 3 mm, malposition and/or endodontic problem
* Maxillary premolars with gingival recession in the palatal area and/or prosthetic restoration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Graft shrinkage | baseline, 1-, 3-months after FGG surgery
  The shrinkage of the graft area was calculated according to the differences between the graft area at baseline, 1st, 3rd months using ImageJ software.

SECONDARY OUTCOMES:
Keratinized tissue weight gain (KTW) | baseline, 1-, 3-months after FGG surgery
  Alginate impressions of each participants were taken from mandibular teeth and an acrylic stent containing both mandibular canine-canine teeth was prepared. The measurements were made relatively with reference to the predetermined points on the stent. KTW was measured as the distance from the buccal midpoint of tooth between the free gingival margin and the alveolar mucosa.

OTHER OUTCOMES:
Relative vestibule depth (rVD) | baseline, 1-, 3-months after FGG surgery
  Alginate impressions of each participants were taken from mandibular teeth and an acrylic stent containing both mandibular canine-canine teeth was prepared. The measurements were made relatively with reference to the predetermined points on the stent. The distance between the reference point on the acrylic stent and mucogingival junction was considered as the relative vestibular depth.
Probing pocket depth (PD) | baseline, 1-, 3-months after FGG surgery
  Probing pocket depth measured as the distance between the base of the pocket and the free gingival margin from the mesial, midbuccal and distal surfaces of the tooth belonging to the surgical site.

CONTACTS AND LOCATIONS:
Overall Officials: Sadiye GUNPINAR, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The authors can share the data upon reasonable request.

REFERENCES:
- [Derived] Shakiliyeva S, Sahin D, Gunpinar S, Gursel M. Comparison of conventional and modified sling suture techniques in free gingival graft operations-a randomized controlled clinical trial. BMC Oral Health. 2025 Feb 21;25(1):279. doi: 10.1186/s12903-025-05456-x. PMID 39984903